CLINICAL TRIAL: NCT03507556
Title: The Regenerative Potential of Immature Necrotic Teeth With Apical Periodontitis Based on Clinical and Radiographic Assessments
Brief Title: Regeneration of Immature Teeth. Case Series
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JordanUST1
Record Dates: First submitted 2018-04-15; First posted 2018-04-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Revascularization
Keywords: immature teeth, necrotic teeth
MeSH Terms: interventions — Zinc Oxide; Ciprofloxacin

STUDY DESIGN:
Intervention Model Description: Revascularization for immature necrotic permanent teeth with apical periodontitis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Triple paste and induced bleeding (Experimental): The triple paste is a mixture of metronidazole, ciprofloxacin and minocycline mixed with sterile glycol will be used and next visit intracanal bleeding will be induced
  Interventions: Procedure: Triple paste and induced bleeding; Drug: Triple Paste metronidazole, ciprofloxacin and minocycline mixed with sterile glycol

INTERVENTIONS:
Procedure: Triple paste and induced bleeding
Drug: Triple Paste metronidazole, ciprofloxacin and minocycline mixed with sterile glycol — triple paste of metronidazole, ciprofloxacin and minocycline mixed with sterile glycol

SUMMARY:
This clinical study aims to investigate the predictability of revascularization procedure of immature necrotic human permanent teeth with apical periodontitis. The quality of root development (thickness and length) will be assessed radiographically.

DETAILED DESCRIPTION:
All teeth will be disinfected using either triple antibiotic paste (a mixture of metronidazole, ciprofloxacin and amoxicillin mixed with sterile glycole) or non setting calcium hydroxide applied to the pulp space with a sterile lentulospiral and then closed temporarily with a sterile sponge and temporary restoration for 2-3 weeks to allow disinfection of the canals teeth will be reentered under rubber dam isolation and all intracanal medicaments will be washed out from the canal using 10 ml of 2.5% sodium hypochlorite and 20 ml of Ethylene diamine tetra acetic acid (EDTA). Then, a sterile endodontic file will be inserted past the canal terminus into the periapical tissues to induce bleeding to fill the canal space as much as possible and subsequently sealed with a double coronal seal using bioceramic repair material and composite filling. All the teeth will be monitored clinically and radiographically on a biannual basis.

ELIGIBILITY:
Inclusion Criteria:

1. Teeth diagnosed with necrotic pulp with/without evidence of apical periodontitis.
2. An immature/open apex.
3. Tooth does not need post and core restoration.
4. Medically healthy patients with no known allergy to used materials.

Exclusion Criteria:

1. Medically compromised patient,
2. Teeth with periodontal involvement
3. Teeth with vertical root fractures,
4. Non-restorable teeth,

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-06-28 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
complete healing | from start of intervention up to 100 months.
  Assess clinically and radiographically absence of symptoms and signs. And evidence for continuation of root development

CONTACTS AND LOCATIONS:
Locations (1):
- Dental health center, Irbid, Jordan